CLINICAL TRIAL: NCT03334331
Title: Validation and Reproducibility of the Six-minute Step Test in Individuals With Obstructive Sleep Apnea Treated With Continuous Positive Airway Pressure (CPAP)
Brief Title: Validation and Reproducibility of the Six-minute Step Test in Individuals With Obstructive Sleep Apnea Treated With CPAP
Status: Completed | Type: Observational
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Matheus Gustavo Silva Magalhães, Principal Investigator, Universidade Federal de Pernambuco
Other Study IDs: 66301817.3.0000.5208
Record Dates: First submitted 2017-10-30; First posted 2017-11-07 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Six-minute step test — Volunteers will be instructed to go up and down one step for six minutes
Other: Six-minute walk test — Volunteers will walk the longest distance possible by performing turns in a 30 meter corridor for six minutes

SUMMARY:
Introduction: The Obstructive Sleep Apnea (OSA) is characterized by obstructed superior airway during sleeping period promoting intermittent hypoxia-reoxygenation events. These events cause consequences such as cardiorespiratory and peripheric muscle structure alterations, which can cause reduction of the exercise tolerance. In this sense the continuous positive airway pressure (CPAP) is important to decrease the repercussions of the illness and cooperate to maintain the exercise functional capacity. To measure this capacity, one good option is the six-minute step test (6MST), that is low cost and submaximal, in addition to being adaptable and portable. However, there are doubts if it´s really capable to determinate the functional capacity of exercise of individuals with OSA treated with CPAP. Objective: Evaluate the validity and reproducibility of 6MST to determine the functional capacity of exercise in individual with OSA treated with CPAP and develop a model of a reference equation for the performance of the test in this population. Material and methods: This is an observational, prospective and cross-sectional study, in which will be evaluated 132 volunteers (66 men and 66 women), with age between 18 and 65 years, diagnosed with OSA of moderate and severe degree, treated with CPAP for a minimum of three months, recruited of the ambulatory of pneumology of Otávio de Freitas Hospital. Initially will be collected personal and anthropometric information, answered to sleep questioners, quality of sleep and physical exercise, also respiratory muscle strength and lung function. The realization of the tests to evaluate the functional capacity of exercise will be done in two days with a maximum of seven days between the tests. In each day, the volunteers will do two 6MST and two six-minute walk test (6MWT), which order will be determined by randomization. Expected Results: It is expected that the 6MST to be showed as reproducible and capable to quantify the functional capability of exercise in individuals with OSA treated with CPAP.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with age between 18 and 65 years;
* Obstructive Sleep Apnea on moderate and severe degree (diagnosed by polysomnography);
* BMI bigger then 18 and less than 35 kg/m2;
* Treatment with CPAP at least three months, with use of the equipment for a time interval superior of 4h/night during five days per week.

Exclusion Criteria:

* Individuals with comorbidities such as uncontrolled hypertension and diabetes, orthopedic and neurologic alterations, respiratory disorders such as COPD and asthma, or any cardiovascular and respiratory which won't permit the realization of the tests.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals adults with obstructive sleep apnea treated with CPAP
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-12-07 (Actual)

PRIMARY OUTCOMES:
Number of steps | Two days
  Number of steps climbed on the six-minute step test
Walked distance | Two days
  Distance walked on six-minute walk test

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Otávio de Freitas, Recife, Pernambuco, Brazil